CLINICAL TRIAL: NCT03763695
Title: Effectiveness of a Bundle of Ventilator Associated Pneumonia (VAP) Prevention in the Pediatric Intensive Care Unit (PICU): an Observational Study
Brief Title: Effectiveness of a VAP Prevention Bundle in the PICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ilaria Vitali (Unknown); Antonio Maria Dell Anna (Unknown); Leonardo Dassatti (Unknown); Giuseppe Bello (Unknown); Giorgio Conti (Unknown); Antonio D Addona (Unknown)
Responsible Party: Principal Investigator, Orazio Genovese, Medical Doctor, pediatric intensive care unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1855
Record Dates: First submitted 2018-09-18; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Pediatric intensive care unit; Oral Hygiene Care; Chlorhexidine; Broncho-alveolar lavage; Pharyngeal swab
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective control group: Patients admitted in our PICU before the implementation of the protocol for VAP prevention (from 01/01/2016 to 12/31/2017)
  Interventions: Other: Evaluation of VAP incidence before the protocol introduction
- Prospective group: Patients admitted to our PICU since the VAP bundle has been introduced in the clinical practice (from 01/01/2018)
  Interventions: Other: Measures for the VAP prevention in the PICU

INTERVENTIONS:
Other: Measures for the VAP prevention in the PICU — Oral hygiene care (i.e chlorhexidine swab); clean and dry ventilator circuits; head positioning at 45 degrees.
  Groups: Prospective group
Other: Evaluation of VAP incidence before the protocol introduction — evaluation of VAP incidence in our pediatric population of intensive care patients before the implementation of the protocol for VAP prevention
  Groups: Retrospective control group

SUMMARY:
This observational monocentric prospective study aims to evaluate the efficacy of new measures for ventilator associated pneumonia (VAP) management in the pediatric population in the pediatric intensive care unit (PICU) of Fondazione Policlinico Agostino Gemelli of 8 beds. The investigators will compare the incidence of VAP in the group of patients in which this protocol has been implemented to a retrospective control group of patients before the new protocol implementation. VAP bundle includes oral care hygiene measures (i.e chlorhexidine swab), to keep clean and dry ventilator circuits and head positioning at 45 degrees.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years
* patients receiving mechanical ventilation for more than 48 hours

Exclusion Criteria:

* no informed consent
* pregnancy
* previous endotracheal antibiotic therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to our ICU requiring mechanical ventilation for more than 48 hours
Sampling Method: Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
VAP incidence | From 48 hours after intubation to 48 hours after extubation
  Incidence of VAP in pediatric patients intubated for more than 48 hours

SECONDARY OUTCOMES:
Prevalence of orotracheal bacterial colonization in ventilated patients | From 48 hours after intubation to 48 hours after extubation
  Evaluation of orotracheal bacterial colonization in pediatric patients undergoing mechanical ventilation twice a week

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Conti, MD, Study Chair — Università Cattolica del Sacro Cuore; Fondazione Policlinico Universitario Agostino Gemelli; IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided